CLINICAL TRIAL: NCT01125397
Title: The Potential Effectiveness of Behavior Therapy on Weight Loss Following Bariatric Surgery
Brief Title: Behavior Therapy Prior to Bariatric Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Karen Grothe, Karen Grothe, PhD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-007135; FP00054166
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: bariatric surgery; behavioral weight management; psychosocial outcomes following bariatric surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Intervention (Experimental)
  Interventions: Behavioral: LEARN group
- Control (No Intervention): These participants will be randomized to receive no behavioral intervention prior to bariatric surgery.

INTERVENTIONS:
Behavioral: LEARN group — Participants will complete a 12-week behavioral weight management intervention (the LEARN program) prior to bariatric surgery, which is the current standard clinical practice at Mayo Clinic Rochester. This involves weekly group meetings, weigh-ins, and goal setting.
  Arms: Behavioral Intervention

SUMMARY:
Obesity is an ever increasing public health problem in this country. Bariatric surgery is currently the most effective treatment for morbid obesity and two hundred thousand surgeries are performed in the United States each year. Unfortunately, despite anatomically successful surgery, it is estimated that at most surgical centers about 30 percent of patients will not achieve significant weight loss following surgery. It has been proposed that participation in preoperative behavior therapy can enhance postoperative outcomes, although empirical evidence for this premise is lacking. The current study is a pilot project designed to conduct a prospective randomized trial to examine the impact of participation in a 12-week standardized preoperative behavioral weight management program on percentage of excess weight loss and psychosocial and medical outcomes at six months after roux-en-Y gastric bypass surgery. The cost of bariatric surgery is not covered by this study and only patients local to the Rochester, Minnesota area are eligible to participate.

It is hypothesized that patients who complete the 12-week behavioral program will experience greater weight loss and improved psychosocial and medical outcomes compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 40 and 60
* age 25 to 65
* ability to participate in weekly LEARN groups for 3 months at Mayo Clinic (local to the Rochester, MN area)
* seeking RYGB procedure

Exclusion Criteria:

* patients seeking surgical revision of a previous bariatric procedure
* diagnosis of schizophrenia
* diagnosis of bipolar disorder
* diagnosis of borderline personality disorder
* non-local patients

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Percent excess weight loss following bariatric surgery | 6 months post-surgery
  The study will compare percent excess weight loss between the two groups (behavioral intervention vs. control)

SECONDARY OUTCOMES:
Psychosocial outcomes | 6 months post-surgery
  Psychological outcomes that will be assessed at baseline and 6 months postoperatively include quality of life (SF-36), depression (BDI-II, PHQ-9), anxiety (GAD-7), alcohol use (AUDIT), distress tolerance (DTS), emotional eating (EOQ), and eating self-efficacy (WEL). All questionnaires are validated and possess good psychometric properties. All measures except the SF-36 are currently given as routine practice during psychological evaluations of bariatric patients, enhancing feasibility for the current study.
Resolution of medical comorbidities | 6 months post-surgery
  Resolution rates of comorbidities will be assessed 6 months post-surgery defined as follows: diabetes as no longer requiring medication and A1C level <7, hypertension as no longer requiring medication and blood pressure of <140 mm Hg (systolic)/90 mm Hg (diastolic). Patients are typically seen at 2 and 6 weeks postoperatively in the surgery clinic and 3 and 6 months in Endocrinology, therefore percentage of follow-up will be calculated as appointments attended/appointments scheduled. Time from initial evaluation until surgery will also be assessed as a possible covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Karen B Grothe, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States